CLINICAL TRIAL: NCT01957397
Title: Investigation of Three Newly Developed 2-piece Convex Base-plates in Subjects With Ileostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP230
Record Dates: First submitted 2013-10-01; First posted 2013-10-08 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coloplast Test 1 (Experimental): The subjects are randomised to two arms
  In both arms the subjects start measuring the performance of own product to collect baseline data.
  In this arm the subjects are randomised to test Coloplast Test1 first and thereafter Coloplast Test 2
  Finally the all subject test Coloplast Test 3
  Interventions: Device: Coloplast Test 1; Device: Coloplast Test 2; Device: Coloplast Test 3
- Coloplast Test 2 (Experimental): The subjects are randomised to two arms
  In both arms the subjects start measuring the performance of own product to collect baseline data.
  In this arm the subjects are randomised to test Coloplast Test 2 first and thereafter Coloplast Test 1
  Finally the all subject test Coloplast Test 3
  Interventions: Device: Coloplast Test 1; Device: Coloplast Test 2; Device: Coloplast Test 3

INTERVENTIONS:
Device: Coloplast Test 1 — Coloplast Test 1 is a newly developed 2-piece convex ostomy appliance
Device: Coloplast Test 2 — Coloplast Test 2 is a newly developed 2-piece convex ostomy appliance
Device: Coloplast Test 3 — Coloplast Test 3 is a newly developed 2-piece convex ostomy appliance

SUMMARY:
To investigate the performance and safety of the three 2-piece convex ostomy appliances

ELIGIBILITY:
Inclusion Criteria:

Subjects interested in participating in the clinical investigation must comply with the following criteria:

1. Are at least 18 years of age and have full legal capacity
2. Have had an ileostomy for at least 3 months.
3. Have used a convex ostomy appliance for the last month
4. Have given written informed consent
5. Have an ileostomy with a diameter of 33mm or less
6. Have experienced leakage (seeping) under the baseplate at least two times over the last two weeks

Exclusion Criteria:

Subjects complying with the following criteria must be excluded from participation in the clinical investigation:

1. Have a loop ostomy (also called double-barrel or ostomy with two outlets)
2. Are pregnant* or breastfeeding.
3. Currently receiving, or have received within the last 2 months, chemotherapy or radiation therapy.
4. Currently receiving or have received, within the last month, systemic or local steroid treatment (adrenocortical hormone) in the peristomal area.
5. Currently suffering from peristomal skin problems (i.e. bleeding or broken skin (weeping skin)).
6. Known hypersensitivity toward any of the test products

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakobsen, MD, Principal Investigator — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects are recruited from the Coloplast A/S user database in Denmark.
Pre-assignment Details: The subjects are randomised to two arms
  In both arms the subjects start measuring the performance of own product to collect baseline data.
  In this arm the subjects are randomised between Coloplast Test1 and Coloplast Test 2
  In the third test period all subject test Coloplast Test 3
Groups:
- 1st Coloplast Test 1,2nd Coloplast Test 2 3rd Coloplast Test 3: The subjects are randomised to two arms
  In both arms the subjects start measuring the performance of own product to collect baseline data.
  In this arm the subjects are randomised to test Coloplast Test1 first and thereafter Coloplast Test 2
  Finally the all subject test Coloplast Test 3
  Coloplast Test 1: Coloplast Test 1 is a newly developed 2-piece convex ostomy appliance
  Coloplast Test 2: Coloplast Test 2 is a newly developed 2-piece convex ostomy appliance
  Coloplast Test 3: Coloplast Test 3 is a newly developed 2-piece convex ostomy appliance
- 1st Coloplast Test 2 2nd Coloplast Test 1 3rd Coloplast Test 3: The subjects are randomised to two arms
  In both arms the subjects start measuring the performance of own product to collect baseline data.
  In this arm the subjects are randomised to test Coloplast Test 2 first and thereafter Coloplast Test 1
  Finally the all subject test Coloplast Test 3
  Coloplast Test 1: Coloplast Test 1 is a newly developed 2-piece convex ostomy appliance
  Coloplast Test 2: Coloplast Test 2 is a newly developed 2-piece convex ostomy appliance
  Coloplast Test 3: Coloplast Test 3 is a newly developed 2-piece convex ostomy appliance
Period: Baseline Own Product
Arm/Group | 1st Coloplast Test 1,2nd Coloplast Test 2 3rd Coloplast Test 3 | 1st Coloplast Test 2 2nd Coloplast Test 1 3rd Coloplast Test 3
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Test Period 1
Arm/Group | 1st Coloplast Test 1,2nd Coloplast Test 2 3rd Coloplast Test 3 | 1st Coloplast Test 2 2nd Coloplast Test 1 3rd Coloplast Test 3
Started | 13 | 13
Completed | 11 | 12
Not Completed | 2 | 1
Not completed — sudden leakage/small bag | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Test Period 2
Arm/Group | 1st Coloplast Test 1,2nd Coloplast Test 2 3rd Coloplast Test 3 | 1st Coloplast Test 2 2nd Coloplast Test 1 3rd Coloplast Test 3
Started | 11 | 12
Completed | 11 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Test Period 3
Arm/Group | 1st Coloplast Test 1,2nd Coloplast Test 2 3rd Coloplast Test 3 | 1st Coloplast Test 2 2nd Coloplast Test 1 3rd Coloplast Test 3
Started | 11 | 11
Completed | 9 | 9
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 2
Not completed — the adhesive did not work | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Population
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage
Description: The degree of leakage was measured with a 32 -point scale developed by Coloplast A/S, where 0 is the best possible outcome (no leakage) and 32 is the worst possible outcome (full leakage under the baseplate)
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: baseplates
Groups:
- Coloplast Test 1: The subjects are randomised to two arms
  In both arms the subjects start measuring the performance of own product to collect baseline data.
  In this arm the subjects are randomised to test Coloplast Test1 first and thereafter Coloplast Test 2
  Finally the all subject test Coloplast Test 3
  Coloplast Test 1: Coloplast Test 1 is a newly developed 2-piece convex ostomy appliance
  Coloplast Test 2: Coloplast Test 2 is a newly developed 2-piece convex ostomy appliance
  Coloplast Test 3: Coloplast Test 3 is a newly developed 2-piece convex ostomy appliance
- Coloplast Test 2: The subjects are randomised to two arms
  In both arms the subjects start measuring the performance of own product to collect baseline data.
  In this arm the subjects are randomised to test Coloplast Test 2 first and thereafter Coloplast Test 1
  Finally the all subject test Coloplast Test 3
  Coloplast Test 1: Coloplast Test 1 is a newly developed 2-piece convex ostomy appliance
  Coloplast Test 2: Coloplast Test 2 is a newly developed 2-piece convex ostomy appliance
  Coloplast Test 3: Coloplast Test 3 is a newly developed 2-piece convex ostomy appliance
- Baseline - Own Product: The subjects test own product to measure their baseline leakage
Arm/Group | Coloplast Test 1 | Coloplast Test 2 | Coloplast Test 3 | Baseline - Own Product
Number analyzed (Participants) | 25 | 24 | 22 | 26
Number analyzed (baseplates) | 146 | 146 | 118 | 166
units on a scale | 4.5 (4.9) | 5.2 (4.8) | 6.4 (5.5) | 6.8 (6.0)

ADVERSE EVENTS:
Time Frame: October - December 2012
Arm/Group | Coloplast Test 1 | Coloplast Test 2 | Coloplast Test 3 | Baseline - Own Product
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/24 | 0/22 | 1/26
Other Adverse Events (participants affected / at risk) | 7/25 | 15/24 | 12/22 | 3/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test 1 (N=25) | Coloplast Test 2 (N=24) | Coloplast Test 3 (N=22) | Baseline - Own Product (N=26)
Expantion of rectal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — The Serious adverse event was not related to the test product
Heart spams (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The serious adverse event was not related to own product
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test 1 (N=25) | Coloplast Test 2 (N=24) | Coloplast Test 3 (N=22) | Baseline - Own Product (N=26)
skin irritation (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (8) | 7 (7) | 1 (1)
Itching of peristomal skin (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 3 (3) | 0 (0)
Pain in the peristomal skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Broken skin in peristomal area (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes